CLINICAL TRIAL: NCT07189767
Title: The Effect of a Psychoeducation Program Applied to Pregnant Women With Traumatic Birth Perception on Maternal Attachment, Breastfeeding, and Postpartum Depression Levels
Brief Title: Effects of Psychoeducation on Pregnant Women With Traumatic Birth Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burcu Firat (Other)
Responsible Party: Sponsor-Investigator, Burcu Firat, Assistant Professor, Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IUC-FNHF-BF-01
Record Dates: First submitted 2025-08-14; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Perception of Traumatic Birth
Keywords: traumatic birth; psychoeducation; perception of birth
MeSH Terms: conditions — Birth Injuries

STUDY DESIGN:
Intervention Model Description: psychoeducation and control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation (Experimental): Pregnant women with a traumatic perception of birth who received psychoeducational intervention formed the experimental group.
  Interventions: Behavioral: psychoeducation
- Control (No Intervention): Pregnant women with a traumatic birth perception who did not receive psychoeducation intervention and underwent routine prenatal follow-up constituted the control group.

INTERVENTIONS:
Behavioral: psychoeducation — The nurse/midwife-led psychoeducation intervention aims to encourage pregnant women to express their feelings about childbirth. It also provides a counseling framework to help women identify and overcome the distressing elements of childbirth. Psychoeducation allows pregnant women to obtain complete, evidence-based information about labor and to discuss their feelings and thoughts about the method of delivery and birth. Providing evidence-based information by nurses/midwives during psychoeducation helps pregnant women make informed decisions about their birth preferences. In addition to evidence-based information, the psychoeducation intervention includes discussing myths and misconceptions, increasing social support, reinforcing positive coping strategies, and focusing on problem solutions. Nurses/midwives encourage pregnant women to develop a positive birth plan through psychoeducation.
  Arms: Psychoeducation

SUMMARY:
The aim of this study is to evaluate the effects of a prenatal psychoeducation program applied to pregnant women with a traumatic perception of birth on the perception of traumatic birth, maternal attachment, breastfeeding and postpartum depression.

DETAILED DESCRIPTION:
Pregnancy and birth are one of the most important experiences in a woman's life. This experience has many physical, hormonal and psychosocial effects on women. The perception of birth varies depending on the culture in which women live. In most societies, birth and motherhood are perceived positively. While some women perceive the experience of giving birth as a positive life experience that strengthens them and helps them grow, some women perceive it as trauma.

The perception of traumatic birth negatively affects the health of mother and baby during pregnancy, birth and the postpartum period. The perception of trauma towards birth causes stress and anxiety disorders, fear of birth, weakening of the bond between mother and baby and the relationship between spouses during pregnancy. During the birth process, it paves the way for increased medical interventions, prolonged labor, decreased success of labor management, and an increased desire for cesarean section. Postpartum problems include failure to participate in infant care, inadequate breastfeeding, decreased breast milk supply, poor mother-infant bonding, postpartum depression, deterioration in family relationships, reluctance to consider future pregnancy, and a tendency toward cesarean section in subsequent pregnancies Removing the perception of birth as traumatic and establishing a positive perception of it is crucial for maternal and infant health. Support should be provided to women who perceive birth as traumatic with practices that have been successful in preventing negative birth experiences. This support allows for the elimination of potential problems resulting from birth trauma . Psychoeducation is one of the most successful practices that will eliminate the perception of traumatic birth. Psychoeducation is one of the most effective evidence-based practices emerging in both clinical research and community settings. It is an educational intervention that includes disease-specific information as well as techniques for managing the current situation. Its flexibility allows it to be used across a wide range of illnesses and life challenges. Studies show that psychoeducation intervention reduces pain levels during labor, increases vaginal birth rates, shortens labor duration, positively affects mother-baby bonding and breastfeeding, and reduces postpartum depression rates.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida
* Between 22 and 32 weeks gestation
* Experiencing a healthy pregnancy
* Spontaneously pregnant
* No psychiatric illness
* Scored 79 or higher on the Traumatic Birth Perception Scale were included in the study.

Exclusion Criteria:

* High-risk pregnant women
* Without a smartphone, tablet, computer or internet access

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 80 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Traumatic Birth Perception Scale (TBPS) | 4 months
  The TBPS was developed in 2016 by Yalnız et al. to determine the level of perception of labor as trauma. The TPAS is used to determine the perceptions of birth among women aged 15-49, receiving preconception counseling, and attending delivery rooms, obstetrics, or postpartum services during pregnancy. The TPAS has a total of 13 items. Each item is rated from 0 (zero) to 10 (ten). The lowest score on the TPAS is 0 (zero), and the highest is 130. As the score on the scale increases, the extent to which women perceive birth as trauma increases. Women who score "0-26" on the scale have a very low perception of birth as traumatic, those who score "27-52" have a low perception, those who score "53-78" have a moderate perception, those who score "79-109" have a high perception, and those who score "105-130" have a very high perception of birth as traumatic. The Cronbach alpha coefficient of the original form of the scale is 0.895.

SECONDARY OUTCOMES:
Mother-to-Infant Bonding Scale (MIBS) | 4 months
  Developed by Taylor and colleagues (2005) to assess mother-infant attachment from the first days after birth to the 12th week, the PBI allows mothers to express their feelings toward their babies in single words after birth. The PBI is a four-point Likert-type scale consisting of 8 items. Each item is scored between 0 and 3. The items cover both positive and negative emotions. Items 1, 4, and 6 examine positive emotions. These items are scored as 0, 1, 2, or 3. Items 2, 3, 5, 7, and 8 examine negative emotions. They are reverse-scored as 3, 2, or 1, or 0. The lowest possible score on the scale is 0, and the highest is 24. A higher score indicates a problem in the mother-infant bond.
Breastfeeding Self-Efficacy Scale Short Form (BSES-SF) | 4 months
  Developed by Dennis and Faux, this scale consists of 14 items on a 5-point Likert-type scale. The lowest possible score is 14, and the highest is 70. A higher score indicates higher breastfeeding self-efficacy. The Turkish validity and reliability of the scale were conducted by Aluş-Tokat and Okumuş (2010).
Edinburgh Postnatal Depression Scale (EPDS) | 4 months
  It was developed by Cox et al. (1987) to determine the risk of depression in mothers during the postpartum period. It consists of 10 items on a 4-point Likert-type scale. The lowest possible score is 0, and the highest is 30. The cut-off point is 12-13. Women who score 13 or higher are at increased risk of postpartum depression. The validity and reliability of the scale in Turkish was conducted by Engindeniz et al. (1996).

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
because there is no release yet

REFERENCES:
- [Background] Pandey Bista A, Shrama C, Shrestha U, Timalsina P, Devkota K, Piya K, Neupane B. Effect of Group Psycho-Educational Interventions on Child birth fear and Child birth Self-efficacy among Primiparous women. J Nepal Health Res Counc. 2023 Jul 20;20(4):846-851. doi: 10.33314/jnhrc.v20i4.4028. PMID 37489666
- [Result] Fenwick J, Toohill J, Gamble J, Creedy DK, Buist A, Turkstra E, Sneddon A, Scuffham PA, Ryding EL. Effects of a midwife psycho-education intervention to reduce childbirth fear on women's birth outcomes and postpartum psychological wellbeing. BMC Pregnancy Childbirth. 2015 Oct 30;15:284. doi: 10.1186/s12884-015-0721-y. PMID 26518597
- [Result] Akgun M, Boz I, Ozer Z. The effect of psychoeducation on fear of childbirth and birth type: systematic review and meta-analysis. J Psychosom Obstet Gynaecol. 2020 Dec;41(4):253-265. doi: 10.1080/0167482X.2019.1689950. Epub 2019 Nov 13. PMID 31718369
- [Result] Boz I, Akgun M, Duman F. A feasibility study of a psychoeducation intervention based on Human Caring Theory in nulliparous women with fear of childbirth. J Psychosom Obstet Gynaecol. 2021 Dec;42(4):300-312. doi: 10.1080/0167482X.2020.1752173. Epub 2020 Apr 22. PMID 32319341
- [Result] Gultekin, N. (2018). Does Psychoeducation Encourage Pregnant Women and Positively Influence the Relation between Mother and Baby: a Case-Control Study. Int J Gynecol Clin Pract, 5(143), 2
- [Result] Jiao N, Zhu L, Chong YS, Chan WS, Luo N, Wang W, Hu R, Chan YH, He HG. Web-based versus home-based postnatal psychoeducational interventions for first-time mothers: A randomised controlled trial. Int J Nurs Stud. 2019 Nov;99:103385. doi: 10.1016/j.ijnurstu.2019.07.002. Epub 2019 Jul 21. PMID 31442783
- [Result] Kordi, M., Bakhshi, M., Masoudi, S., & Esmaily, H. (2017). Effect of a childbirth psychoeducation program on the level of fear of childbirth in primigravid women. Evidence Based Care, 7(3), 26-34.
- [Result] Lawrence CG, Breau G, Yang L, Hellerstein OS, Hippman C, Kennedy AL, Ryan D, Shulman B, Brotto LA. Effectiveness of a web-enabled psychoeducational resource for postpartum depression and anxiety among women in British Columbia. Arch Womens Ment Health. 2024 Dec;27(6):995-1010. doi: 10.1007/s00737-024-01468-8. Epub 2024 May 6. PMID 38709329
- [Result] Maharani Dewi, U., Windarti, Y., & Hayani, H. (2023). The Effect of Lactation Psychoeducation Using a Video-Based Comprehensive Model on the Level of Anxiety of Mothers in Breastfeeding. Health Education and Health Promotion, 11(3), 1001-1013.
- [Result] Hollander MH, van Hastenberg E, van Dillen J, van Pampus MG, de Miranda E, Stramrood CAI. Preventing traumatic childbirth experiences: 2192 women's perceptions and views. Arch Womens Ment Health. 2017 Aug;20(4):515-523. doi: 10.1007/s00737-017-0729-6. Epub 2017 May 29. PMID 28553692
- [Result] Firouzan L, Kharaghani R, Zenoozian S, Moloodi R, Jafari E. The effect of midwifery led counseling based on Gamble's approach on childbirth fear and self-efficacy in nulligravida women. BMC Pregnancy Childbirth. 2020 Sep 9;20(1):522. doi: 10.1186/s12884-020-03230-1. PMID 32907547
- [Result] Fenwick J, Toohill J, Slavin V, Creedy DK, Gamble J. Improving psychoeducation for women fearful of childbirth: Evaluation of a research translation project. Women Birth. 2018 Feb;31(1):1-9. doi: 10.1016/j.wombi.2017.06.004. Epub 2017 Jul 3. PMID 28684046
- [Result] Kuipers YJ, Thomson G, Goberna-Tricas J, Zurera A, Hresanova E, Temesgenova N, Waldner I, Leinweber J. The social conception of space of birth narrated by women with negative and traumatic birth experiences. Women Birth. 2023 Feb;36(1):e78-e85. doi: 10.1016/j.wombi.2022.04.013. Epub 2022 May 2. PMID 35514007
- [Result] Nagle U, Naughton S, Ayers S, Cooley S, Duffy RM, Dikmen-Yildiz P. A survey of perceived traumatic birth experiences in an Irish maternity sample - prevalence, risk factors and follow up. Midwifery. 2022 Oct;113:103419. doi: 10.1016/j.midw.2022.103419. Epub 2022 Jul 9. PMID 35930929